CLINICAL TRIAL: NCT06118658
Title: A Single-arm, Open, Multicenter Phase II Study of Chemotherapy-sequential Tislelizumab Adjuvant Therapy After Radical Resection in Patients With Gastric or Colorectal Adenocarcinoma With dMMR/MSI-H or POLE/POLD1 Mutations
Brief Title: Chemotherapy Sequential Tislelizumab After Radical Resection in Patients With dMMR/MSI-H or POLE/POLD1 Mutations
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Jingdong Zhang, Chief physician, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adjuvant-GC/EGJ/CRC
Record Dates: First submitted 2023-10-29; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Gastric; Colorectal Adenocarcinoma
Keywords: radical resection; adjuvant therapy; gastric; colorectal adenocarcinoma; esophagogastric junction adenocarcinoma; dMMR/MSI-H or POLE/POLD1 mutations
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: About 30 patients who underwent radical gastrectomy or enterectomy with gastric adenocarcinoma or esophagogastric junction adenocarcinoma with postoperative pathological stage III or intestinal adenocarcinoma with postoperative pathological stage T1-3N2M0 or T4N+M0(American Joint Committee on Cancer,AJCC 8th Edition Cancer Stage) were scheduled to be enrolled after fully informed and signed informed consent Qualified subjects were selected to receive the standard XELOX or SOX regimen selected by the investigators according to the disease and postoperative pathology of the subjects for 4 cycles, followed by the sequential treatment of monotherapy tislelizumab (200mg,Q3W, IV infusion,4 cycles) starting from 4-6 weeks after surgery, with a maximum of 12 weeks Safety assessments such as ECOG physical examination of vital signs and laboratory tests will be performed regularly during treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy-sequential tislelizumab adjuvant therapy (Experimental): About 30 patients who underwent radical gastrectomy or enterectomy with gastric adenocarcinoma or esophagogastric junction adenocarcinoma with postoperative pathological stage III or intestinal adenocarcinoma with postoperative pathological stage T1-3N2M0 or T4N+M0(American Joint Committee on Cancer,AJCC 8th Edition Cancer Stage) were scheduled to be enrolled after fully informed and signed informed consent Qualified subjects were selected to receive the standard XELOX or SOX regimen selected by the investigators according to the disease and postoperative pathology of the subjects for 4 cycles, followed by the sequential treatment of monotherapy tislelizumab (200mg,Q3W, IV infusion,4 cycles) starting from 4-6 weeks after surgery, with a maximum of 12 weeks Safety assessments such as ECOG physical examination of vital signs and laboratory tests will be performed regularly during treatment
  Interventions: Drug: tislelizumab

INTERVENTIONS:
Drug: tislelizumab — About 30 patients who underwent radical gastrectomy or enterectomy with gastric adenocarcinoma or esophagogastric junction adenocarcinoma with postoperative pathological stage III or intestinal adenocarcinoma with postoperative pathological stage T1-3N2M0 or T4N+M0(American Joint Committee on Cancer,AJCC 8th Edition Cancer Stage) were scheduled to be enrolled after fully informed and signed informed consent Qualified subjects were selected to receive the standard XELOX or SOX regimen selected by the investigators according to the disease and postoperative pathology of the subjects for 4 cycles, followed by the sequential treatment of monotherapy tislelizumab (200mg,Q3W, IV infusion,4 cycles) starting from 4-6 weeks after surgery, with a maximum of 12 weeks Safety assessments such as ECOG physical examination of vital signs and laboratory tests will be performed regularly during treatment

SUMMARY:
Objective of this study to evaluate 1-year disease-free survival in patients with dMMR/MSI-H or POLE/POLD1 gene mutations with gastric or esophagus-gastric junctional adenocarcinoma or colorectal adenocarcinoma after chemotherapy-sequential tiralizumab adjuvant radical resection (based on RECIST v1.1 criteria).

DETAILED DESCRIPTION:
Colorectal cancer and gastric cancer are common malignant tumors of digestive tract. The latest statistical data show that the number of new cases of colorectal cancer and gastric cancer in China ranks second and third among all malignant tumors, and the number of death cases ranks fifth and third. They are one of the main cancers threatening the life and health of Chinese residents, causing serious social burden In recent years, immunotherapy represented by immune check point inhibitors (ICI) has made great progress in the treatment of malignant tumors, among which programmed death receptor 1(pro grammed death) 1,PD-1) antibody is the most widely used.

Microsatellite instablehigh (MSI-H) is highly unstable due to DNA mismatch repairdeficient (dMMR) .The insertion or loss of the base pairs of microsatellite fragments, the change of the length of microsatellite tandem repeats, and the emergence of new microsatellite alleles are one of the mechanisms of tumor occurrence. Deficient mismatch repair (dMMR)/ microsatellite instablehigh (MSI-H) is the first molecular marker discovered to predict the efficacy of ICI treatment for pancancer .The emergence of ICI therapy has brought the dawn for prolonging the survival time of patients with advanced gastrointestinal tumors.Immune checkpoint inhibitors have shown satisfactory results in patients with MSI-H/dMMR from late-stage to first-line therapy.A 2015 study by Le et al.was the first to show that molecular phenotypic metastatic colorectal (mCRC) with mismatch repair defects (dMMR) or high microsatellite instability (MSI-H) can benefit significantly from the immune checkpoint PD-1 inhibitor pembrolizumab. Immune checkpoint inhibitors have made significant progress in the treatment of the posterior line of colorectal cancer.In KEYMAT-016, a pivotal study of MSI-H tumor immunotherapy, multiple tumors of dMMR benefited from PD-1 monoclonal antibody Pbolizumab. For mCRC patients who failed standard therapy, 7 out of 13 dMMR/MSI-H patients received pembrolizumab monotherapy and achieved objective remission (62%) .All patients did not achieve median progression-free time (PFS) and overall survival time (OS), and the KEYNOTE-164 study further investigated dMMR/MSI-H The clinical benefit of pabolizumab in mCRC patients was an objective response rate (ORR) of 32%(median follow-up 12.6 months) and 1-year progression-free survival and overall survival were 41% 76%, respectively, among 63 previously treated patients in KEYMAT-164 Cohort B This study shows that MSI-H CRC patients treated with pabolizumab have sustained anti-tumor effects even after first-line therapy progresses.The KEYNOTE-059 trial, which included patients with metastatic gastric/gastroesophageal junction tumors after second-line chemotherapy failure, showed an ORR of 47%(3/7) in the MSI-H group compared to only 9%(15/167) in the non-MSI-H group.In KEYNOTE 158, the ORR for MSI-H gastric cancer treated with pembrolizumab reached 45.8% (11/24 95% CI: 25.6% ~ 67.2%) .A number of subgroup analyses have shown that MSI-H gastric cancer has advantages over chemotherapy in immunotherapy, and adverse drug reactions are within the acceptable range. A number of PD-1/PD-L1 models have been approved for the treatment of unresectable or metastatic MSI-H/dMMR solid tumors. Immune checkpoint inhibitors not only show surprising efficacy in the posterior treatment of patients with advanced tumors, but also have been confirmed as first-line treatment. CheckMate142、KEYNOTE-177 study explored the efficacy of immunotherapy as first-line treatment of bowel cancer, and both achieved promising OS and PFS results.KEYNOTE-177 MSI-H first-line patients treated with pembrolizumab for advanced colorectal cancer significantly extended median PFS(16.5 months vs.8.2 months) and improved ORR(43.8%vs.33.1%) compared to standard chemotherapy. This study also established the position of immunotherapy in the first-line treatment of MSI-H advanced colorectal cancer, further supporting the gradual push of immunotherapy from the back line treatment to the front line treatment.

However, the role of immunotherapy in the adjuvant treatment of MSI-H/dMMR solid tumors is still uncertain. No matter NCCN guidelines, ESMO guidelines or China's CSCO guidelines, for postoperative adjuvant treatment of people with advantages of immune benefit, observation or chemotherapy is recommended according to the stage and risk factors. Based on the remarkable results achieved in previous studies, the role of immunotherapy in MSI-H/dMMR adjuvant therapy for colon and gastric cancer is worthy of expectation.

tislelizumab is a humanized IgG4 anti-PD-1 monoclonal antibody, which is currently the only PD-1 antibody modified by Fc segment. It removes the binding ability of FC-γR on the surface of macrophages, does not mediate the cross-linking of immune cells, avoids the ADCP effect to the greatest extent, avoids T cell consumption, and theoretically enhances its anti-tumor activity. RATIONALE 209 study results show that patients with MSI-H metastatic solid tumor who failed standard therapy receiving tislelizumab monotherapy can also achieve an impressive objective response rate (ORR(mCRC :39%; G/GEJC :55.6%), the security is controllable. tislelizumab has been approved by NMPA for the treatment of urothelial carcinoma, non-small cell lung cancer, hepatocellular carcinoma, esophageal squamous cell carcinoma, nasopharyngeal carcinoma, and highly microsatellite unstable solid tumors.

POLE/POLD1 mutations encoding DNA polymerase are involved in the occurrence and development of various tumors, and the mutation rate of POLE/POLD1 is about 7.4% in colorectal cancer and 7.1% in esophageal cancer. Mutations in the gene encoding POLE and POLD1 exonuclide region lead to loss of correction function, which is closely related to tumor hypermutation, TMB elevation, neogenic antigen increase, and increased intra tumor immune cell infiltration. Previous studies have shown that these are closely related to good immune efficacy, which also indicates that POLE/POLD1 mutation is expected to become a molecular marker for predicting the efficacy of ICI, a new pan-cancer species.

In summary,MSI-H/dMMR and POLE/POLD1 mutations are advantageous populations for immunotherapy. The purpose of this study was to explore the efficacy and safety of chemotherapy followed by tislelizumab for adjuvant treatment of gastric or esophago-gastric junctional adenocarcinoma or colorectal adenocarcinoma in patients with radical resection of dMMR/MSI-H or POLE/POLD1 mutations. To provide clinical guidance for MSI-H/dMMR or POLE/POLD1 gene mutated colon and gastric cancer adjuvant therapy modalities

ELIGIBILITY:
Inclusion Criteria:

1.Be able to understand and voluntarily sign a written informed consent, which must be signed prior to performing the specified study procedure required for the study 2.Age and gender: ≥18 years old and≤75 years old, both men and women. 3.dMMR/MSI-H or POLE/POLD1 gene mutation was confirmed by immunohistochemical PCR or NGS 4.0-1 physical fitness score by the Eastern United States Cancer Collaboration (ECOG)。 5. Expected survival is 12 weeks 6.Radical gastrectomy or enterectomy, including open surgery or laparoscopic surgery, to achieve R0 resection (no residual cancer at the margin) 7.According to the American Joint Committee on Cancer AJCC 8th Edition cancer stage, it was confirmed by histopathology as gastric adenocarcinoma or esophagogastric junction adenocarcinoma or intestinal adenocarcinoma, and the postoperative pathological stage of gastric adenocarcinoma or esophagogastric junction adenocarcinoma was stage III; Patients with postoperative pathological stage of intestinal cancer T1-3N2M0 or T4N+M0 8.No metastasis or recurrence was determined based on images taken after surgery and within the first 28 days of randomization 9. Subjects are required to provide sufficient FFPE tumor tissue specimens or sections for relevant testing 10.The functions of important organs must meet the following requirements:

1. Hematological system（No blood component or cell growth factor was used to support treatment within 7 days prior to the start of study therapy）:

   Neutrophil count≥1.5×10^9/L; Platelet count≥100×10^9/L; Hemoglobin≥90g/L;
2. Liver function： Serum albumin≥28g/L; Total bilirubin (TBI)≤1.5×ULN; Alanine aminotransferase (ALT)≤3×ULN Aspartate aminotransferase (AST)≤2.5×ULN
3. Renal function:

   Serum creatinine ≤1.5×ULN Calculated creatinine clearance≥50 mL/min (using the Cockcroft-Gault formula); Female: CrCl = (140- age in years) × weight in kg × 0.85 72 × serum creatinine in mg/ dL

   Male: CrCl = (140- age in years) × weight in kg × 1.00 72 × serum creatinine in mg/ dL
4. Coagulation function:

   Subjects not receiving anticoagulation therapy: INR or APTT ≤ 1.5×ULN;
5. Cardiac function: Left ventricular ejection fraction (LVEF)≥ 50 10. Fertile female subjects must undergo a urine or serum pregnancy test within 3 days prior to the first dosing (if the urine pregnancy test result is not confirmed negative, a serum pregnancy test is required, depending on the serum pregnancy result), and the result is negative If a fertile female subject has sex with an unsterilized male partner, the subject must use a highly effective contraceptive method since screening and must consent to continued use of the contraceptive method for 120 days after the last administration of the study drug; Whether to stop contraception after this time point should be discussed with the investigator 11.If an unsterilized male subject has sex with a fertile female partner, the subject must use an effective contraceptive method from the beginning of screening until the 120th day after the last dose; Whether to stop contraception after this time point should be discussed with the investigator.

12.Subjects were willing and able to comply with the schedule for visiting treatment protocol laboratory tests and other study requirements.

Exclusion Criteria:

1. Subjects with other malignancies in the 5 years prior to enrolment do not exclude subjects with other malignancies that have been cured by local treatment, such as basal or skin squamous cell carcinoma superficial bladder cancer cervix or breast carcinoma in situ
2. Have received non-surgical treatment for gastric/esophagogastric junction/bowel cancer (e.g., radiotherapy, chemotherapy and hormone therapy)
3. Liver peritoneum or distant metastasis
4. Inability to take medications orally
5. Unrelieved postoperative complications during screening (such as postoperative infection, suture rupture, gastrointestinal bleeding, pancreatic leakage, etc.)
6. There are chemotherapy drugs contraindicated in this study and any group of adjuvant therapy regiments specified in the regimen cannot be accepted
7. People with active autoimmune diseases that have required systemic treatment within the past two years (such as treatment with disease-modifying drugs, corticosteroids, immunosuppressants) and replacement therapy (such as insulin thyroxine or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) are not considered a systemic treatment
8. There is a pleural, pericardial or abdominal effusion that is clinically symptomatic, requires diuretic treatment and/or requires repeated drainage.
9. There are active or recurrent inflammatory gastrointestinal diseases (such as Crohn's disease ulcerative colitis hemorrhagic enteritis chronic diarrhea, etc.)
10. A history of myocarditis and cardiomyopathy with malignant arrhythmias.Unstable angina pectoris, myocardial infarction, congestive heart failure (grade 2 or higher according to the New York Heart Association Functional Scale), or vascular disease (such as an aortic aneurysm at risk of rupture) requiring hospitalization in the 12 months prior to initial administration,Or other heart damage that may affect the safety evaluation of the investigational drug (e.g., poorly controlled arrhythmias, myocardial ischemia)
11. Medically difficult to control hypertension (systolic blood pressure ≥150mmHg and/or diastolic blood pressure ≥100mmHg) (based on an average of ≥2 measurements).
12. Uncontrolled diabetes.
13. Peripheral neuropathy ≥ grade 2.
14. Severe infection within 4 weeks prior to initial dosing, including but not limited to comorbidized sepsis or severe pneumonia requiring hospitalization; Active infections that have received systemic anti-infective therapy within 2 weeks prior to initial dosing (excluding antiviral therapy for hepatitis B or C)
15. Known active tuberculosis (TB), suspected active TB subjects need to undergo clinical examination to rule out; Known active syphilis infection
16. Subjects with current active hepatitis B (HBsAg positive with more than 2000 copies /ml(500 IU/ml) of HBV-DNA or higher than the lower limit of detection, whichever is higher), for subjects with hepatitis B, are required to receive anti-HBV therapy during the study treatment; Active hepatitis C subjects (HCV antibody positive with HCV-RNA levels above the lower limit of detection)
17. History of immune deficiency; HIV antibody test positive; Systemic corticosteroid hormones or other immunosuppressants are currently being used on a long-term basis
18. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
19. Prior treatment with PD-1 receptor or its ligand PD-L1 or cytotoxic T lymphocyte-associated protein 4(CTLA-4) receptor
20. Known allergy to any component of any investigational drug; There is a known history of severe hypersensitivity to other monoclonal antibodies
21. Inactivated vaccines are allowed if a live or attenuated vaccine has been administered in the 30 days prior to the first dose, or if a live or attenuated vaccine is planned to be administered during the study
22. Known history of mental illness substance abuse alcohol or drugs
23. Pregnant or lactating women
24. The presence of any past or current abnormality in laboratory tests for treatment of disease that may confuse the study results, affect the subject's full participation in the study, or participation in the study may not be in the subject's best interest
25. Local or systemic disease caused by non-malignant tumors; Or disease or symptoms secondary to the tumor and can lead to higher medical risk and/or uncertainty in the evaluation of survival
26. Any condition that the investigator believes may cause subjects to receive the study drug treatment to be at risk of interfering with the evaluation of the study drug, or affecting the interpretation of the study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year disease-free survival based on RECIST v1.1 criteria (1-year DFS rate) | 1-year
  The 1-year DFS rate was defined as the proportion of all subjects who did not have disease recurrence within 1 year from the start of randomization.

SECONDARY OUTCOMES:
1-year MRD-negative survival assessed based on MRD testing | 1 year
  Proportion of all subjects tested MRD negative at 1 year from randomization.
Disease-free survival (DFS) | DFS is defined as the time from the start of randomization until a subject's disease recurrences or death from any cause, whichever occurs first
  DFS is defined as the time from the start of randomization until a subject's disease recurrences or death from any cause, whichever occurs first
overall survival (OS) | OS is defined as the time from randomization to death from any cause
  OS is defined as the time from randomization to death from any cause
time to local recurrence (TTLR) | TTLR was defined as the time from randomization to local tumor recurrence.
  TTLR was defined as the time from randomization to local tumor recurrence.
time to recurrence (TTR) | TTR is defined as the time from randomization to tumor recurrence (including local recurrence and distant metastasis).
  TTR is defined as the time from randomization to tumor recurrence (including local recurrence and distant metastasis).

OTHER OUTCOMES:
dMMR/MSI-H POLE/POLD1 gene mutation, TMB and its dynamic changes, and the relationship between efficacy and adverse reactions | Subject recurrence of disease or discontinuation of treatment for any reason
  dMMR/MSI-H POLE/POLD1 gene mutation, TMB and its dynamic changes, and the relationship between efficacy and adverse reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Liaoning Cancer Hospital & Institute, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No